CLINICAL TRIAL: NCT02572596
Title: A Prospective Control Study of Comparing Intermediate-dose Cyclophosphamide(ID-CTX) and G-CSF Plus or Not Recombinant Human Thrombopoietin (rhTPO) for PBSC Mobilization in Patients With Multiple Myeloma
Brief Title: Comparing Intermediate-dose CTX+ G-CSF Plus or Not rhTPO for PB CD34+ Cells Mobilization in MM Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wang Guorong (Other)
Responsible Party: Sponsor-Investigator, Wang Guorong, Clinical Professor, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MM-TPO-01
Record Dates: First submitted 2015-09-17; First posted 2015-10-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Multiple Myeloma
Keywords: Hematopoietic Stem Cell Mobilization; Thrombopoietin
MeSH Terms: conditions — Multiple Myeloma; Jacobs syndrome | interventions — Thrombopoietin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhTPO treatment group (Experimental): Subject will receive chemotherapy with intermediate-dose CTX 2.5/m2 for 2 days. 10 ug/kg/d of G-CSFwas administered from the WBC was lower than 1×10^9/L following bejing of chemotherapy or no later than day 7after chemotherapy. G-CSF was subcutaneously administered once daily until the stem cell collection was completed. rhTPO was administered 15 000 U/d once daily by subcutaneous injection from day 5-7 after chemotherapy and until the stem cell collection was completed.
  Interventions: Drug: rhTPO; Drug: CTX; Drug: -CSF
- non- rhTPO treatment group (Active Comparator): Subject will receive chemotherapy with intermediate-dose CTX 2.5/m2 for 2 days. 10 ug/kg/d of G-CSF was administered from the WBC was lower than 1×10^9/L following bejing of chemotherapy or no later than day 7after chemotherapy. G-CSF was subcutaneously administered once daily until the stem cell collection was completed.
  Interventions: Drug: CTX; Drug: -CSF

INTERVENTIONS:
Drug: rhTPO — rhTPO was administered 15 000 U/d once daily by subcutaneous injection from day 5-7 after chemotherapy and until the stem cell collection was completed.
  Other Names: recombinant human thrombopoietin; Recombinant Human TPO
  Arms: rhTPO treatment group
Drug: CTX — CTX 2.5/m2 for 2 days.
  Other Names: Cyclophosphamide
Drug: -CSF — 10 ug/kg/d of G-CSFwas administered from the WBC was lower than 1×10^9/L following bejing of chemotherapy or no later than day 7after chemotherapy. G-CSF was subcutaneously administered once daily until the stem cell collection was completed.
  Other Names: granulocyte colony-stimulatingG

SUMMARY:
Comparing intermediate-dose CTX (ID-CTX)and G-CSF with rhTPO or without for peripheral blood stem cell mobilization in patients with multiple myeloma, try to find out whether rhTPO combined to ID-CTX + G-CSF could improve the results of peripheral blood stem cell mobilization.

DETAILED DESCRIPTION:
The purpose of this study is to try to find out whether rhTPO combined to ID-CTX + G-CSF could improve the results of peripheral blood stem cell mobilization. Comparing ID-CTX and G-CSF plus rhTPO or not for peripheral blood stem cell mobilization in patients with multiple myeloma. rhTPO15000U/d were given from day 5~7 after chemotherapy until the stem cell collection .

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed MM fulfill the International Myeloma Working Group (IMWG) criteria for MM diagnosis
* Eastern Cooperative Oncology Group (ECOG) performance status smaller than 2 and a life expectancy of more than 6 months
* Age at least 18 ys , no more than 70 ys old
* No active infectious disease; no severe organ failure (except renal failure secondary to MM)
* All screening procedures and evaluations should be completed
* All patients should provide written informed consent.

Exclusion Criteria:

1. severe impaired liver function; HIV positive or had active hepatitis A, B or C infection; hepatitis B virus-DNA more than 10^4/L;aspartate aminotransferase ( AST) and alanine aminotransferase (ALT) more than 2.5 upper limit of normal (ULN)
2. any disease that could put patients at high risk, including but not limited to unstable cardiac disease, defined as myocardial infarction in the previous 6 months, New York Heart Association (NYHA) class III-IV heart failure, uncontrolled atrial fibrillation or hypertension
3. severe prior thrombosis-event
4. history of other malignancy, unless cured for more than 3 years
5. pregnancy, lactation or disagreement to take contraceptive measures
6. severe infectious disease (uncured tuberculosis, pulmonary aspergillosis)
7. epilepsia, dementia or any mental disease requiring treatment.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2013-01-01; Primary Completion 2017-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of CD34+ stem/progenitor cells that are mobilized | two weeks

SECONDARY OUTCOMES:
rate of mobilization success | two weeks
rate of mobilization optimal | two weeks

OTHER OUTCOMES:
occurrence rate of febrile neutropenia | three weeks
platelet transfusion amount | three weeks
time of neutrophil engraftment | four weeks
time of platelet engraftment | eight weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Chen, doctor, Principal Investigator — Beijing Chao Yang Hospital,CCMU
Locations (1):
- Beijing Chaoyang Hospital, Beijing, Beijing Municipality, China